CLINICAL TRIAL: NCT05589571
Title: An Evaluation of the Relationship Between Physiological Parameters of Stress and In Vitro Fertilization Outcome
Brief Title: Evaluation of the Impact of Stress on IVF Outcome
Status: Completed | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: OTO US Fertility LP (Unknown)
Responsible Party: Sponsor
Other Study IDs: INC-2022-002
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Stress, Physiological; Infertility; Stress, Psychological
Keywords: IVF; In-vitro fertilization; OTO; Inception; Stress; Omegawave; Infertility; FET; Frozen embryo transfer
MeSH Terms: conditions — Infertility; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine if physiological measures of stress, measured by the non-invasive OTO device, are significantly correlated with IVF outcome.

DETAILED DESCRIPTION:
The OTO device is a wearable device that utilizes multiple methods of electrophysiology to identify the impact of stress on humans. The device consists of the OTO sensor, a belt with two electrode pads worn around the chest, one electrode placed on the thenar of the dominant hand and one electrode placed on the forehead; the sensor pairs with the OTO App via Bluetooth. It tracks 54 physiological properties including temperature, HRV, amplitude frequency analysis (AFA) of ECG and DC potential. This data is analyzed by the proprietary OTO Expert System which creates the overall conclusions on levels of stress, functional reserves, adaptive capacity and level of readiness to additional stressors.

Physiological data will be collected from the study participant using the OTO device for the duration of one IVF and frozen embryo transfer (FET) cycle. Study participants will complete questionnaires online related to perceived stress at the beginning and the end of study participation. Study participant's IVF cycle treatment and outcome data will be collected and analyzed in conjunction with the physiological data collected with the OTO device.

ELIGIBILITY:
Inclusion Criteria:

* Women age 25-40 years old
* Planning to undergo their first IVF cycle with frozen embryo transfer at one of the participating fertility clinics
* Have access to the internet and own a smartphone
* Ability and willingness to wear the OTO device for a few minutes each morning during their IVF and FET cycle
* Able to read and speak English

Exclusion Criteria:

* Medical history of cardiac arrhythmias
* History of cardiac surgery within a year of study enrollment

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between age 25-40 years old who are scheduled to undergo their first IVF and frozen embryo transfer cycle at one of the participating fertility clinics.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Physiological Stress | 7 weeks
  Physiological stress will be measured using the non-invasive OTO device, which tracks 54 physiological properties including temperature, hear rate variability (HRV), amplitude frequency analysis (AFA) of electrocardiogram (ECG) and direct current (DC) potential.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Domar, PhD, Principal Investigator — Inception Fertility Research Institute, LLC
Locations (42):
- United States (42):
  - IVFMD, Boca Raton, Florida
  - Center for Reproductive Medicine, Celebration, Florida
  - IVFMD, Cooper City, Florida
  - IVFMD, Jupiter, Florida
  - IVFMD, Miami, Florida
  - IVFMD, Naples, Florida
  - IVFMD, Viera, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Reproductive Biology Associates, Atlanta, Georgia
  - Reproductive Biology Associates, Cumming, Georgia
  - Reproductive Biology Associates, Lawrenceville, Georgia
  - Reproductive Biology Associates, Marietta, Georgia
  - Advanced Fertility Center of Chicago, Chicago, Illinois
  - Advanced Fertility Center of Chicago, Crystal Lake, Illinois
  - Advanced Fertility Center of Chicago, Downers Grove, Illinois
  - Advanced Fertility Center of Chicago, Gurnee, Illinois
  - Indiana Fertility Institute, Indianapolis, Indiana
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - Main Line Fertility, Havertown, Pennsylvania
  - Main Line Fertility, Paoli, Pennsylvania
  - Main Line Fertility, Philadelphia, Pennsylvania
  - Main Line Fertility, West Chester, Pennsylvania
  - Tennessee Fertility Institute, Franklin, Tennessee
  - Tennessee Fertility Institute, Nashville, Tennessee
  - Aspire Fertility Austin, Austin, Texas
  - Aspire Houston Fertility Institute, Beaumont, Texas
  - Aspire Houston Fertility Institute, Cypress, Texas
  - Aspire Fertility Dallas, Dallas, Texas
  - Aspire Houston Fertility Institute - Memorial City, Houston, Texas
  - Aspire Houston Fertility Institute - Main Street, Houston, Texas
  - Aspire Houston Fertility Institute - Medical Center, Houston, Texas
  - Aspire Houston Fertility Institute - Piney Point, Houston, Texas
  - Aspire Houston Fertility Institute - Willowbrook, Houston, Texas
  - Aspire Houston Fertility Institute, Katy, Texas
  - Aspire Houston Fertility Institute, Kingwood, Texas
  - Aspire Fertility McAllen, McAllen, Texas
  - Aspire Houston Fertility Institute, Pearland, Texas
  - Aspire Fertility San Antonio - Medical Center, San Antonio, Texas
  - Aspire Fertility San Antonio - Sonterra, San Antonio, Texas
  - Aspire Houston Fertility Institute, Sugar Land, Texas
  - Aspire Houston Fertility Institute, The Woodlands, Texas
  - Aspire Houston Fertility Institute, Webster, Texas

REFERENCES:
- See also: Inception Network Fertility Studies - OTO — http://fertilitystudies.com/oto/